CLINICAL TRIAL: NCT05666414
Title: Assessment of Vertical Bone Gain and Neurosensory Affection in Computer Guided vs Conventional Sandwich Osteotomy Technique in the Atrophied Posterior Mandible: a Randomized Clinical Trial
Brief Title: Vertical Bone Gain and Neurosensory Affection in Computer Guided vs Conventional Sandwich Osteotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Khaled Mohamed, teaching assisstant, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: (24)/11-2021
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer guided sandwich interpositional bone grafting (Experimental): patient specific cutting guide were fabricated to perform the osteotomies ( and another patient specific guide was then fabricated to start the fixation of the cut bony segment a full digital intervention for sandwich interpositional grafting in patients with vertically atrophied mandible (bilateral split mouth study)
  Interventions: Procedure: sandwich interpositional bone grafting computer guided
- conventional sandwich osteotomy interpositional bone grafting (Active Comparator): conventional interpositional bone grafting was done for patients with vertically atrophied mandibles (bilateral split mouth study)
  Interventions: Procedure: conventional interpositional bone grafting

INTERVENTIONS:
Procedure: sandwich interpositional bone grafting computer guided — performing the 2 vertical and the 1 horizontal osteotomies using a cutting patient specific guide and fixation of the vertically elevated bony segment after gap calculation using patient specific fixation guides
  Arms: computer guided sandwich interpositional bone grafting
Procedure: conventional interpositional bone grafting — performing the conventional interpositional sandwich osteotomies free-hand and fixation of the mobilized bone segment free-hand
  Arms: conventional sandwich osteotomy interpositional bone grafting

SUMMARY:
The aim of this study was to assess the efficiency of the computer-guided interpositional sandwich osteotomy for the vertical bone gain and effects on vital structures (inferior dental nerve bundle) compared to free hand interpositional osteotomies.

DETAILED DESCRIPTION:
in this research a full digital sandwich osteotomy protocol was conducted to be compared with the conventional protocol. the investigators were seeking to determine the significance of using surgical computer software in sandwich interpositional bone grafting at atrophied posterior mandibles and how efficiently can it affect this technique.

ELIGIBILITY:
Inclusion Criteria:

* • Edentulous posterior mandibular ridge with vertical loss of alveolar bone with remaining bone height (4-7 mm) above the mandibular canal

  * Good oral hygiene
  * Highly motivated patients
  * Patients seeking fixed prosthesis at posterior mandibular region.
  * Patients willing for a surgical procedures follow-up with an informed consent
  * Age range 20-65 years

Exclusion Criteria:

* • Smokers

  * Individuals with dentulous posterior mandible ridge
  * Medically compromised patients
  * Patients with local pathosis at the surgical area suggested
  * Previously subjected to reconstructive procedures of the posterior mandible

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
amount of vertical bone gain | 4 months
  measure the amount of vertical bone gained after performing the interpositional sandwich osteotomy

SECONDARY OUTCOMES:
neurosensory affection | 4 months
  measure the affection of the inferior alveolar nerve bundle after performing the interpositional sandwich osteotomy

CONTACTS AND LOCATIONS:
Overall Officials: ahmed k mohamed, BDS, Principal Investigator — university
Locations (1):
- Future University in Egypt, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No